CLINICAL TRIAL: NCT02823730
Title: Registry Experience at the Washington Hospital Center With Drug Eluting Stents - Synergy (REWARDS-Synergy)
Brief Title: Registry Experience at the Washington Hospital Center With Drug Eluting Stents - Synergy
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REWARDS-Synergy
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Incidence of Major Adverse Cardiac Events

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Synergy Stent Cohort: Retrospective registry of 500 patients who have received the Synergy stent. Data will be mined from the DES registry database for the identified Synergy patients at the following time points, in-hospital and then at 1 year, 2 years, 3 years, and 4 years after percutaneous coronary intervention (PCI).
  Interventions: Other: PCI with Synergy Stent
- Xience V Cohort: 500 patients that are propensity matched to the 500 patients that underwent PCI with a Synergy stent, eligible for similar time points of follow-up following the PCI.

INTERVENTIONS:
Other: PCI with Synergy Stent — 500 patients who have received the Synergy stent. Data will be mined from the DES registry database for the identified Synergy patients at the following time points, in-hospital and then at 1 year, 2 years, 3 years, and 4 years after percutaneous coronary intervention (PCI).
  Groups: Synergy Stent Cohort

SUMMARY:
To compare the incidence of major adverse cardiac events among a series of patients receiving the Synergy drug-eluting stent with bioabsorbable polymer to historical controls who have received the Promus Premier drug-eluting stent with durable polymer.

DETAILED DESCRIPTION:
The primary objective of this observational, real-world single-center registry is to compare the incidence of major adverse cardiac events among a series of patients receiving the Synergy drug-eluting stent with bioabsorbable polymer to historical controls who have received the Promus Premier drug-eluting stent with durable polymer. The investigators hypothesize that the long-term incidence (each year following implantation, up to 4 years) of major adverse cardiovascular events, after propensity matching for stent type, will be similar between Synergy and Xience V.

ELIGIBILITY:
Inclusion Criteria:

1. Subject >18 years of age
2. Underwent PCI with Synergy (alone) DES

Exclusion Criteria:

1. Underwent PCI with a non-Synergy DES (or scaffold) during the same index procedure
2. Patients not taking, or unable to take, dual antiplatelet therapy (DAPT) at the time of screening for the study (patients that discontinue DAPT after enrollment will be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center, observational, retrospective registry of 500 patients who have received the Synergy stent. Data will be mined from the DES registry database for the identified Synergy patients at the following time points, in-hospital and then at 1 year, 2 years, 3 years, and 4 years after percutaneous coronary intervention (PCI).
  The 500 patients that underwent PCI with a Synergy stent will then be compared to a propensity matched Xience V cohort eligible for similar time points of follow up following the PCI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 4 years
  major adverse cardiac events (MACE), defined as the composite of: 1. All-cause death; 2. Q-wave myocardial infarction (QwMI): appearance of new pathologic Q waves in the coronary distribution of the target vessel with an increase of creatine kinase-MB to ≥2 times the reference values (if available); 3. Target vessel revascularization (TVR): need for repeat PCI within the target vessel.

SECONDARY OUTCOMES:
Target lesion revascularization | 4 years
  Need for repeat PCI within the target lesion
Periprocedural creatine kinase-MB | 4 years
  peak level of in-hospital CK-MB post-PCI
Cardiac death | 4 years
  Any death due to a cardiovascular cause
Stent thrombosis | 4 years
  Probable or definite stent thrombosis occurring in the target vessel.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States